CLINICAL TRIAL: NCT04695925
Title: A Phase III, Multicentre, Randomized Controlled Study Comparing Osimertinib Monotherapy to Combination Therapy With Osimertinib, Carboplatin and Pemetrexed for Untreated Patients With Advanced Nonsquamous Non-Small Cell Lung Cancer With Concurrent EGFR and TP53 Mutations(TOP)
Brief Title: Osimertinib Monotherapy or Combination With Chemotherapy for Advanced NSCLC Concurrent EGFR and TP53 Mutations
Acronym: TOP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Li Zhang, MD (Other)
Collaborators: Cancer Hospital of Guangxi Medical University (Other); First People's Hospital of Foshan (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Li Zhang, MD, Principal Investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21647
Record Dates: First submitted 2020-12-20; First posted 2021-01-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Carcinoma; EGFR Gene Mutation
MeSH Terms: interventions — osimertinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- osimertinib monotherapy (Active Comparator): Osimertinib, 80mg, QD, p.o. until disease progression
  Interventions: Drug: Osimertinib
- combination of osimertinib and chemotherapy (Experimental): Osimertinib, 80mg, QD, p.o. Pemetrexed 500 mg/m2 and carboplatin area under curve 5 intravenously every 3 weeks for four cycles, followed by maintenance pemetrexed.
  Interventions: Drug: Osimertinib; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Osimertinib — Osimertinib, 80mg, QD, p.o. until disease progression
Drug: Pemetrexed — pemetrexed 500 mg/m2 intravenously every 3 weeks until disease progression
  Arms: combination of osimertinib and chemotherapy
Drug: Carboplatin — carboplatin area under curve 5 intravenously every 3 weeks for four cycles
  Arms: combination of osimertinib and chemotherapy

SUMMARY:
This is a phase III randomized trial in patients with advanced non-squamous NSCLC harboring EGFR-sensitizing mutations and concurrent TP53 mutations with a performance status of 0 to1 who are planned to receive first-line therapy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label, phase III study comparing the progression free survival, overall survival, response rate, toxicity, quality of life between Osimertinib monotherapy and combination of osimertinib, pemetrexed, carboplatin in first-line treatment of advanced non-small cell lung cancer patients with concurrent EGFR and TP53 mutation. Besides, the association between other genetic mutations and efficacy will also be analyzed as exploratory endpoint. Eligible patients will be randomized to receive either osimertinib or osimertinib combined with pemetrexed and carboplatin in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Male or female, aged at least 18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1;
4. Life expectancy of at least 3 months;
5. Histologically or cytologically confirmed stage IV or recurrent non-squamous non-small cell lung carcinoma with activating EGFR mutations (exon 19 deletion or exon 21 L858R point mutation) and concurrent TP53 mutations;
6. No prior palliative chemotherapy, or palliative biological (including targeted therapies such as EGFR and vascular epidermal growth factor (VGEF) inhibitors) or immunological therapy （Previous adjuvant chemotherapy is permitted if treatment was completed more than 6 months before day 1. Palliative radiotherapy to a metastatic site is permitted, but palliative wide field radiotherapy to the lung must be completed at least 4 weeks before day 1 with no persistence of any radiotherapy-related toxicity;
7. Adequate organ function, including the following:

   * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) counts (ANC) ≥ 1.5X109/L, Platelets ≥100X109/L, HGB ≥90g/L. The use of granulocyte colony stimulating factor support, platelet transfusion and blood transfusions to meet these criteria is not permitted;
   * Tumour Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (x ULN) if no liver metastases or ≤ 3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases; alanine aminotransferase (ALT) & aspartate aminotransferase (AST) ≤ 2.5 x ULN if no demonstrable liver metastases or AST&ALT ≤ 5 x ULN in the presence of liver metastases;
   * Serum Creatinine ≤ 1.5 times the ULN and Creatinine Clearance ≥ 50 ml/min.
8. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening
9. Post-menopausal defined as aged 50 years or more and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
10. Women under 50 years old would be consider postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site);
2. Previous randomization in the present study or previous treatment with Osimertinib;
3. Known severe hypersensitivity to Osimertinib or any of the excipients of this product;
4. Known severe hypersensitivity to carboplatin, pemetrexed or any of the excipients of these products;
5. Known severe hypersensitivity to pre-medications required for treatment with carboplatin/ pemetrexed doublet chemotherapy;
6. History or presence of any other malignancy with the exception of basal cell carcinoma or cervical cancer in situ;
7. Past medical history of interstitial lung disease, drug induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease;
8. Any unresolved chronic toxicity ≥ CTCAE grade 2 from previous anticancer therapy;
9. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease);
10. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study;
11. Pregnancy or breast feeding;
12. Use of unapproved drugs or research drugs within 30 days before the start of the study;
13. Symptomatic brain metastases.
14. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value;
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block;
    * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes;
    * Correction of electrolyte abnormalities to within normal ranges can be performed during screening;
15. Pre-existing idiopathic pulmonary fibrosis evidence by CT scan at baseline;
16. Unable to tolerate carboplatin/pemetrexed doublet chemotherapy, as judged by the investigator;
17. Life expectancy of ≤ 12 weeks;
18. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection (e.g. patients receiving treatment for infection) including hepatitis C and human immunodeficiency virus (HIV), or active uncontrolled HBV infection;
19. Screening for chronic conditions is not required. Should participants with HBV infection be included, patients are only eligible if they meet all the following criteria:

    * Demonstrated absence of HCV co-infection or history of HCV co-infection;
    * Demonstrated absence of HIV infection;
    * Participants with active HBV infection are eligible if they are: Receiving anti-viral treatment for at least 6 weeks prior to study treatment, HBV DNA is suppressed to <100 IU/mL and transaminase levels are below ULN;
    * Participants with a resolved or chronic infection HBV are eligible if they are:
    * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG]. In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (TBD by hepatologist) post treatment or
    * Positive for HBsAg, but for >6 months have had transaminases levels below ULN and HBV DNA levels below<100 IU/mL (i.e., are in an inactive carrier state). In addition, patients must be receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (TBD by hepatologist) post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | assessed up to 36 months
  defined as the time from randomization to the date of first documentation of from date of randomization until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
overall survival | OS maturity reaches 60%, assessed up to 60 months
  from date of randomization until the date of death from any cause
percentage of participants with objective response (partial response [PR] plus complete response [CR]) | up to 36 months
  assessed using RECIST v.1.1
Incidence and severity of adverse events (AEs) | through study completion, an average of 60 months
  Overall incidence of AEs; the incidence of grade 3 or above AEs; the incidence of severe adverse events (SAE); the incidence of drug-related AEs; the incidence of AEs resulting in permanent withdrawal of drugs; the incidence of AEs leading to dose adjustment
Change from baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) Score. | up to 36 weeks
  The EORTC QLQ-C30 consists of 30 questions that comprise aspects of participant's functioning assessment (physical, emotional, role, cognitive, and social); symptom scales (fatigue; nausea, vomiting, and pain; the global health/quality of life [QoL]); and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties), within a recall period of "the past week." Most questions used a 4-point scale (1=Not at all to 4=Very much; two questions used a 7-point scale (1=Very poor to 7=Excellent). Scores were averaged and transformed to a 0-100 scale; a higher score for Global Qol/functional scales=better level of functioning; a higher score for symptom scale=greater degree of symptoms.

OTHER OUTCOMES:
Correlation between subtypes of EGFR mutations, TP53 mutations and other potential predictive biomarkers and response to treatment. | up to 36 months
  We do next generation sequencing in tumor tissue and blood sample to detect EGFR, TP53 and additional mutations in other oncogenic drivers and tumor-suppressor genes at baseline. NGS in blood sample is required at the first efficacy assessment (6th week). Upon PD, NGS in blood sample is required while in tumor tissue is preferred.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Medical Oncology,Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong
  - Central Hospital of Guangdong Nongken, Zhanjiang Cancer Hospital, Zhanjiang

IPD SHARING:
Plan to Share IPD: No